CLINICAL TRIAL: NCT05959213
Title: Preoperative CA 19.9 Level Predicts Lymph Node Metastasis in Resectable Adenocarcinoma of the Head of the Pancreas: a Further Plea for Biological Resectability Criteria.
Brief Title: Preoperative CA 19.9 Level Predicts Lymph Node Metastasis in Resectable Adenocarcinoma of the Head of the Pancreas.
Acronym: ICALYRA
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Campus Bio-Medico (Other)
Responsible Party: Principal Investigator, Tommaso Farolfi, Principal investigator, Fondazione Policlinico Universitario Campus Bio-Medico
Other Study IDs: FPUCampusBioMedico
Record Dates: First submitted 2023-05-23; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Pancreas Cancer
Keywords: Ca 19.9; Pancreatic adenocarcinoma; Pancreatoduodenectomy
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In our multicenter retrospective study, preoperative CA 19.9 levels predicts the presence of lymph node metastasis at final histology in patients underwent pancreatoduodenectomy for pancreatic ductal adenocarcinoma .

DETAILED DESCRIPTION:
A retrospective analysis have been conducted on more than 2.000 patients underwent pancreatoduodenectomy for pancreatic ductal adenocarcinoma radiologically resectable at the preoperative staging. Preoperatory levels of CA 19.9 were measured in order to identify a relation with nodal involvement at the pathological staging.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergone pancreatoduodenectomy
* No preoperative radiological suspicion of lymph node metastases.

Exclusion Criteria:

- Age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 2,034 patients were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 2034 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Quantitative data - Preoperatory levels of CA 19.9 (U/ml) | 20 years
  Define relation of quantitative data (CA 19.9 (U/ml)) with nodal positivity at the final pathological report

IPD SHARING:
Plan to Share IPD: No
Upon reasonable request to the Investigator